CLINICAL TRIAL: NCT03806101
Title: A PHASE 1, RANDOMIZED, 2-WAY CROSSOVER, MULTIPLE-DOSE, OPEN-LABEL STUDY TO ESTIMATE THE EFFECT OF PF-04965842 ON ROSUVASTATIN PHARMACOKINETICS IN HEALTHY PARTICIPANTS
Brief Title: Study of PF-04965842 Effect on Rosuvastatin Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B7451033; 2018-003425-28 (EudraCT Number); DDI (Other: Alias Study Number)
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Healthy
MeSH Terms: interventions — abrocitinib; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Single dose of rosuvastatin on Day 1 of Period 1 and Single dose of rosuvastatin on Day 1 + PF-04965842 on Days 1 to 3 of Period 2.
  Interventions: Drug: PF-04965842; Drug: Rosuvastatin
- Arm 2 (Experimental): Single dose of rosuvastatin on Day 1 + PF-04965842 on Days 1 to 3 of Period 1 and single dose of rosuvastatin on Day 1 of Period 2.
  Interventions: Drug: PF-04965842; Drug: Rosuvastatin

INTERVENTIONS:
Drug: PF-04965842 — 200 mg dose of PF-04965842 once daily (QD) for 3 days
Drug: Rosuvastatin — Single 10 mg dose of rosuvastatin

SUMMARY:
This is a Phase 1, randomized, 2 way crossover, multiple dose, open label study of the effect of PF 04965842 on rosuvastatin PK in healthy participants. Participants will be randomized to 1 of the 2 treatment sequences. A total of approximately 12 healthy male and/or female participants will be enrolled in the study so that approximately 6 participants will be enrolled in each treatment sequence. Each treatment sequence will consist of 2 periods. In both sequences, participants will remain in the CRU for a total of 11 days and 10 nights (including Period 1 and Period 2). To adequately remove any drug effects of rosuvastatin from Period 1 to Period 2, there will be a minimum 5 day washout period between the 2 rosuvastatin dosing events.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Age and Sex:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).

   Type of Participant and Disease Characteristics:
2. Male and female participants who are overtly healthy as determined by medical evaluation including a detailed medical history, complete physical examination, laboratory tests, and ECG.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

   Weight:
4. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

   Informed Consent:
5. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic (including alcoholic liver disease, nonalcoholic steatohepatitis (NASH), autoimmune hepatitis, and hereditary liver diseases), psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Evidence of acute exacerbation or history of clinically significant dermatological condition (eg, contact dermatitis or psoriasis) or visible rash present during physical examination.
3. Participants, who according to the product label for rosuvastatin, would be at increased risk if dosed with rosuvastatin.
4. Self reported history or risk factors for QT prolongation or torsades de pointes (eg, organic heart disease, congestive heart failure, hypokalemia, hypomagnesaemia, congenital long QT syndrome, myocardial ischemia or infarction), congenital deafness, family history of sudden death, and family history of long QT syndrome.
5. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, appendectomy).
6. A current or past medical history of conditions associated with thrombocytopenia, coagulopathy or platelet dysfunction.
7. History of human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus infection; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb). As an exception, a positive hepatitis B surface antibody (HepBsAb) as a result of participant vaccination is permissible.
8. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

Prior/Concomitant Therapy:

10. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product.

10. Use of CYP2C19 inhibitors (eg, fluconazole, fluoxetine, fluvoxamine, ticlopidine omeprazole, voriconazole, cimetidine, esomeprazole, and felbamate) or inducers (eg, rifampin, ritonavir, efavirenz, enzalutamide, phenytoin, and St. John's Wort) within 28 days or 5 half-lives (whichever is longer) prior to dosing.

11. Use of CYP2C9 inhibitors (eg, amiodarone, felbamate, fluconazole, miconazole, piperine, diosmin, disulfiram, fluvastatin, fluvoxamine, voriconazole, efavirenz, isoniazid) or inducers (eg, aprepitant, carbamazepine, enzalutamide, rifampin, ritonavir, nevirapine, phenobarbital, and St. John's Wort) within 28 days or 5 half lives (whichever is longer) prior to dosing.

12. Use of CYP3A4 inhibitors (eg, ketoconazole, ciprofloxacin, diltiazem) or other inducers (eg, phenytoin, carbamazepine) within 28 days or 5 half-lives (whichever is longer) prior to dosing.

Prior/Concurrent Clinical Study Experience:

13. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product used in this study (whichever is longer).

Diagnostic Assessments:

14. A positive urine drug test. 15. Screening supine systolic blood pressure (BP) <90 mm Hg or >=140 mm Hg following at least 5 minutes of supine rest; OR Screening supine diastolic BP <50 mm Hg or >=90 mm Hg following at least 5 minutes of supine rest.

If a participant meets any of these criteria, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.

16. Screening supine 12 lead ECG demonstrating:

* QTcF >450 msec; OR
* QRS interval >120 msec. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility.

  17. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:
* Alkaline phosphatase, creatine kinase, aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) level > ULN.
* Total bilirubin level > ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <=ULN.
* Estimated creatinine clearance <90 mL/min.
* Confirmed microscopic proteinuria or hematuria.

Other Exclusions:

18. History of regular alcohol consumption exceeding 14 drinks per week for female participants or 21 drinks per week for male participants (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.

19. Known relevant history of elevated liver function tests (LFTs). 20. History of tuberculosis (TB) (active or latent) or inadequately treated TB infection. Positive QuantiFERON - TB Gold test.

21. Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of baseline.

22. History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.

23. History of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or considered clinically significant by the investigator within 6 months prior to screening.

24. History of receiving a live vaccine within 6 weeks prior to the first dose of investigational product, or is expected to receive a live vaccine within 6 weeks after the last dose of investigational product.

25. Have a known immunodeficiency disorder or a first-degree relative with a hereditary immunodeficiency.

26. History of sensitivity to heparin or heparin induced thrombocytopenia. 27. Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.

28. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to first dose of investigational product.

29. History of hypersensitivity to rosuvastatin. 30. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.

31. Have any malignancies or have a history of malignancies with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.

32. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
AUCinf of rosuvastatin. | 72 hrs after rosuvastatin administration in Period 1 and 2
  Area under the curve from time zero to extrapolated infinite time for rosuvastatin
CLr of rosuvastatin | 72 hrs after rosuvastatin administration in Period 1 and 2
  Renal clearance for rosuvastatin

SECONDARY OUTCOMES:
AUClast of rosuvastatin | 72 hours after rosuvastatin administration in Period 1 and 2
  Area under the plasma concentration time curve from 0 to the time of last measurement of rosuvastatin
Tmax of rosuvastatin | 72 hours after rosuvastatin administration in Period 1 and 2
  Time to maximum concentration of rosuvastatin
Cmax of rosuvastatin | 72 hours after rosuvastatin administration in Period 1 and 2
  Maximum observed plasma concentration for rosuvastatin
t1/2 of rosuvastatin | 72 hours after rosuvastatin administration in Period 1 and 2
  apparent terminal half life of rosuvastatin
Ae of rosuvastatin | 72 hours after rosuvastatin administration in Period 1 and 2
  Amount of rosuvastatin excreted in urine
Ae% of rosuvastatin | 72 hours after rosuvastatin administration in Period 1 and 2
  Percent of dose of rosuvastatin excreted in urine
Number of subjects with adverse events (AEs). | Screening up to 28-35 days after the last dose of PF 04965842 in period 2
  Number of subjects with adverse events (AEs)
Number of subjects with laboratory tests findings of potential clinical importance | Screening through Day 5 of period 2
  Number of subjects with laboratory tests findings of potential clinical importance
Number of subjects with clinically significant abnormal vital signs | Screening through Day 5 of period 2
  Number of subjects with clinically significant abnormal vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Vourvahis M, Byon W, Chang C, Le V, Diehl A, Graham D, Tripathy S, Raha N, Luo L, Mathialagan S, Dowty M, Rodrigues AD, Malhotra B. Evaluation of the Effect of Abrocitinib on Drug Transporters by Integrated Use of Probe Drugs and Endogenous Biomarkers. Clin Pharmacol Ther. 2022 Sep;112(3):665-675. doi: 10.1002/cpt.2594. Epub 2022 May 9. PMID 35344588
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7451033&StudyName=A+Phase+1%2C+Randomized%2C+2-way+Crossover%2C+Multiple-dose%2C+Open-label+Study+To+Estimate+The+Effect+Of+Pf-04965842+On+Rosuvastatin+Pharmacokinetics+In+Healthy+Participants